CLINICAL TRIAL: NCT00347061
Title: A Long-term Safety and Efficacy of SL77.0499-10 10mg Once-daily Tablets in Patients With Lower Urinary Tract Symptoms Related to Benign Prostatic Hyperplasia (BPH).A Multicenter, 52-week, Open Label, Uncontrolled Study.
Brief Title: Long Term Safety of SL77.0499-10 (Alfuzosin) in Patients With BPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS5235
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasiam; Adrenergic alpha-antagonist
MeSH Terms: conditions — Prostatic Hyperplasia

INTERVENTIONS:
Drug: afuzosin

SUMMARY:
Primary:

To assess the safety of SL77.0499-10 10mg administered once daily for one year in patients with lower urinary tract symptoms related to BPH.

Secondary:

* To provide the information on the efficacy of SL77.0499-10 10mg administered once daily for one year in patients with lower urinary tract symptoms related to BPH.
* To document the plasma concentration of SL77.0499-10 after repeated administration of SL77.0499-10 10mg administered once daily in patients with lower urinary tract symptoms related to BPH.

ELIGIBILITY:
Inclusion Criteria:

* Having a symptomatic BPH diagnosed clinically by digital rectal examination and ultrasonography
* Suffering for at least 6 months from lower urinary tract symptoms related to BPH
* An I-PSS total score ≥ 13
* Out patient

Exclusion Criteria:

* Patients previously treated with SL77.0499-10.
* Neurogenic bladder dysfunction, confirmed or suspected, irrespective of aetiology.
* Isolated bladder neck disease.
* Diagnosed carcinoma of the prostate.
* Previous prostatic surgery or other invasive procedures (thermotherapy…) for the treatment of BPH.
* Patients having an indwelling catheter.
* A residual urine > 200mL.
* Patients with Moderate or sever hepatic insufficiency.
* Known hypersensitivity to alpha1-blockers.
* Patients who have received anti-androgens, 5alpha-reductase inhibitors, LH-RH analogues within the previous 3 months before Screening
* Patients judged inappropriate for admission to the study by the Investigator or the Sub-Investigator.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
One year safety data of SL77.0499-10

SECONDARY OUTCOMES:
One year efficacy data and plasma concentration of SL77.0499-10

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan